CLINICAL TRIAL: NCT00418821
Title: A Multicenter, Multinational, Open-Label Study of the Effects of Aldurazyme® (Laronidase) Treatment on Lactation in Women With Mucopolysaccharidosis I (MPS I) and Their Breastfed Infants
Brief Title: A Study of the Effect of Aldurazyme® (Laronidase) Treatment on Lactation in Female Patients With Mucopolysaccharidosis I (MPS I) and Their Breastfed Infants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was conducted to fulfill a post marketing commitment (PMC). FDA acknowledged closure of PMC.
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBS12874; 2007-007003-33 (EudraCT Number); ALID01803 (Other: company study code)
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mucopolysaccharidosis I; Hurler's Syndrome; Hurler-Scheie Syndrome; Scheie
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laronidase (Experimental): Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase and their infants who were breastfeed while the mothers were receiving laronidase.
  Interventions: Biological: Laronidase

INTERVENTIONS:
Biological: Laronidase — dose of 0.58mg/kg body weight intravenously (IV) every week
  Other Names: Aldurazyme; Recombinant human alpha L iduronidase

SUMMARY:
The purpose of this study is to determine if laronidase is present in the breast milk of post-partum women receiving Aldurazyme® (laronidase) and the effects of Aldurazyme (laronidase) on the growth, development, and immunologic response of their breastfed infants.

DETAILED DESCRIPTION:
Recruitment is not limited to the facility listed; facilities not yet active may be added upon identification of a patient.

ELIGIBILITY:
Inclusion Criteria (Mothers):

* The patient must have a documented laronidase deficiency with a fibroblast, plasma, serum, leukocyte, or dried blood spot laronidase enzyme activity assay.
* Be pregnant, planning to breastfeed post-partum, and receiving Aldurazyme (laronidase) therapy while breastfeeding.
* Provide signed, written informed consent prior to any protocol-related procedures. Consent of a legally authorized guardian(s) is (are) required for mothers younger than 18 years of age. If a mother is under 18 years old and can understand the consent, written informed consent is required from both the mother and the authorized guardian(s).
* Provide signed, written informed consent for their infants to participate as study patients. If a mother is younger than 18 years of age, consent for mother and infant will be obtained from the legal guardian.

Exclusion Criteria (Mothers and Infants):

* Have a medical condition, serious intercurrent illness, or other extenuating circumstance that may interfere with study compliance, including all prescribed evaluations and follow-up activities.
* Have received an investigational drug within 30 days prior to study enrollment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-10-22 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Dipartimento di Scienze Pediatriche Medico - Chirurgiche e Neuro Scienze dello Suiluppo, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Castorina M, Antuzzi D, Richards SM, Cox GF, Xue Y. Successful pregnancy and breastfeeding in a woman with mucopolysaccharidosis type I while receiving laronidase enzyme replacement. therapy. Clin Exp Obstet Gynecol. 2015;42(1):108-13. PMID 25864295
- See also: Successful pregnancy and breastfeeding in a woman with mucopolysaccharidosis type I while receiving laronidase enzyme replacement therapy — https://doi.org/10.12891/ceog1845.2015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted to fulfill a post marketing commitment (PMC). Upon acknowledgement of closure of PMC by FDA, the study was terminated by the Sponsor.
Period: Overall Study
Arm/Group | Laronidase
Started | 2
Completed | 1
Not Completed | 1
Not completed — Fulfils one of the exclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Laronidase
Number analyzed (Participants) | 2
Age, Customized [Number; unit: participants]
  Newborns (0-27 days) | 1
  Adults (between 18 and 64 years) | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Based on the low enrolment numbers, no data is reported here in order to protect and maintain participant privacy/confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Number of Lactating Women With Serum IgG Antibodies to Laronidase
Time Frame: Up to 18 months
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Count of Participants; unit: Participants
Groups:
- Laronidase: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase. Mothers received commercially available laronidase as per the country labeling information at the study site.
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Amount of IgG Antibody Titers to Laronidase in Lactating Women
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase
Measure: Mean (Standard Deviation); unit: antibody titer
Groups:
- Laronidase: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Arm/Group | Laronidase
Number analyzed (Participants) | 1
antibody titer
  Baseline | 25600 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 51200 (NA) — Standard deviation cannot be derived for a single participant.

3. Primary Outcome: Number of Women Who Breastfed
Time Frame: Up to 18 months
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants | 1

4. Primary Outcome: Number of Women Who Were Successful at Breastfeeding
Time Frame: Up to 18 months
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants | 1

5. Primary Outcome: Number of Women Whose Breast Milk Contains Laronidase
Time Frame: Up to 18 months
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants | 0

6. Primary Outcome: Amount of Laronidase in the Breast Milk of Lactating Mothers With Mucopolysaccharidosis I (MPS I) Disease
Time Frame: Up to 18 months
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase. There were no women whose breast milk contained laronidase hence overall number of participants analyzed is zero.
Arm/Group | Laronidase
Number analyzed (Participants) | 0

7. Primary Outcome: Number of Women With Abnormal Urine Glycosaminoglycans (uGAG) Levels
Time Frame: Up to 18 months
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants | 0

8. Primary Outcome: Amount of uGAG in the Urine of Women
Description: Urine samples were collected at specified intervals to measure uGAG in the urine of women. Reference range of uGAG between 2.64 - 37.65 was considered as normal. mg/g creatinine = milligram per gram of creatinine.
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Mean (Standard Deviation); unit: mg/g creatinine
Arm/Group | Laronidase
Number analyzed (Participants) | 1
mg/g creatinine
  Baseline | 28.13 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 26.98 (NA) — Standard deviation cannot be derived for a single participant.

9. Primary Outcome: Number of Participants With Medical History of the Mother: Pre-Existing Conditions
Time Frame: Baseline
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants
  Mucopolysaccharidosis type I | 1
  Aortic valvular insufficiency | 1
  Stipsi | 1
  Carpal tunnel syndrome | 1

10. Primary Outcome: Physical Examination Findings of the Mother
Description: Physical examination was performed at specified intervals. Physical examination included the following physical observations: general appearance, skin, head, ears, eyes, nose, and throat, lymph nodes, abdomen, extremities/joints, neurological, mental status, and the following, if appropriate, breasts, external genitalia, pelvic, and rectal.
Time Frame: Up to 18 months
Population: Based on the low enrolment numbers, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Laronidase
Number analyzed (Participants) | 0

11. Primary Outcome: Temperature of the Mother
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase. Temperature was not measured at Week 12.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Celsius
  Baseline | 35.8 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12: number analyzed (Participants) | 0

12. Primary Outcome: Heart Rate of the Mother
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase. Heart rate was not measured at Week 12.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Laronidase
Number analyzed (Participants) | 1
beats per minute
  Baseline | 90 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12: number analyzed (Participants) | 0

13. Primary Outcome: Respiratory Rate of the Mother
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase. Respiratory rate was not measured at Baseline and Week 12.
Arm/Group | Laronidase
Number analyzed (Participants) | 0

14. Primary Outcome: Blood Pressure of the Mother
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured at specified timepoints.
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase. Blood pressure was not measured at Week 12.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Laronidase
Number analyzed (Participants) | 1
millimeters of mercury
  SBP at Baseline | 125 (NA) — Standard deviation cannot be derived for a single participant.
  DBP at Baseline | 80 (NA) — Standard deviation cannot be derived for a single participant.
  SBP at Week 12: number analyzed (Participants) | 0
  DBP at Week 12: number analyzed (Participants) | 0

15. Primary Outcome: Weight of the Mother
Time Frame: Baseline and Week 12
Population: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Laronidase
Number analyzed (Participants) | 1
kilograms
  Baseline | 58.5 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 51 (NA) — Standard deviation cannot be derived for a single participant.

16. Primary Outcome: Height of the Mother
Time Frame: Baseline
Population: as for outcome 10
Arm/Group | Laronidase
Number analyzed (Participants) | 0

17. Primary Outcome: Number of Infants With Abnormal uGAG Levels
Time Frame: Up to 72 weeks
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Count of Participants; unit: Participants
Groups:
- Laronidase: Infants who were breastfeed while the mothers were receiving laronidase.
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants | 1

18. Primary Outcome: Amount of uGAG in the Urine of Infants
Description: Urine samples were collected at specified intervals to measure uGAG in the urine of infant. Reference range of uGAG between 30 - 300 was considered as normal.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, Week 60, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. No sample was collected at Week 60.
Measure: Mean (Standard Deviation); unit: mg/g creatinine
Arm/Group | Laronidase
Number analyzed (Participants) | 1
mg/g creatinine
  Baseline | 76 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 194 (NA) — Standard deviation cannot be derived for a single participant.
  Week 24 | 29 (NA) — Standard deviation cannot be derived for a single participant.
  Week 36 | 55 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 45 (NA) — Standard deviation cannot be derived for a single participant.
  Week 60: number analyzed (Participants) | 0
  Week 72 | 44 (NA) — Standard deviation cannot be derived for a single participant.

19. Primary Outcome: Number of Participants With Medical History of the Infant:Pre-Existing Conditions
Time Frame: Baseline
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants
  Extremities/Joints (clinodactily hands) | 1
  Skin (bilateral transverse palmar crease) | 1

20. Primary Outcome: Number of Infants With Abnormal Physical Finding
Description: Physical examination included the following physical observations: general appearance, skin, lymph nodes, heart, lungs, abdomen, extremities/joints, neurological, mental status, breasts, external genitalia, pelvic, rectal, and Heent.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Number; unit: participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
participants
  Extremities/Joints at Baseline (clinodactily hands) | 1
  Skin at Baseline (bilateral transverse palmar crease) | 1
  Skin at Week 12 (bilateral transverse palmar crease) | 1
  Skin at Week 24 (bilateral transverse palmar crease) | 1
  Skin at Week 36 (bilateral transverse palmar crease almost disappeared) | 1
  Lungs at Week 48 (grunting) | 1
  Skin at Week 72 (bilateral transverse palmar crease) | 1

21. Primary Outcome: Heart Rate of the Infant
Description: Heart rate was measured at specified timepoints.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. Heart rate was not measured at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Laronidase
Number analyzed (Participants) | 1
beats per minute
  Baseline: number analyzed (Participants) | 0
  Week 12 | 121 (NA) — Standard deviation cannot be derived for a single participant.
  Week 24: number analyzed (Participants) | 0
  Week 36 | 102 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 120 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 | 119 (NA) — Standard deviation cannot be derived for a single participant.

22. Primary Outcome: Respiratory Rate of the Infant
Description: Respiratory rate was measured at specified timepoints.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. Respiratory rate was not measured at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Laronidase
Number analyzed (Participants) | 1
breaths/min
  Baseline: number analyzed (Participants) | 0
  Week 12 | 18 (NA) — Standard deviation cannot be derived for a single participant.
  Week 24: number analyzed (Participants) | 0
  Week 36 | 13 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 16 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 | 23 (NA) — Standard deviation cannot be derived for a single participant.

23. Primary Outcome: Blood Pressure of the Infant
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured at specified timepoints.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. Blood pressure was not measured at Baseline, Week 12, and Week 24.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Laronidase
Number analyzed (Participants) | 1
millimeters of mercury
  Baseline SBP: number analyzed (Participants) | 0
  Week 12 SBP: number analyzed (Participants) | 0
  Week 24 SBP: number analyzed (Participants) | 0
  Week 36 SBP | 90 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 SBP | 87 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 SBP | 90 (NA) — Standard deviation cannot be derived for a single participant.
  Baseline DBP: number analyzed (Participants) | 0
  Week 12 DBP: number analyzed (Participants) | 0
  Week 24 DBP: number analyzed (Participants) | 0
  Week 36 DBP | 48 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 DBP | 52 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 DBP | 54 (NA) — Standard deviation cannot be derived for a single participant.

24. Primary Outcome: Weight of the Infant
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Laronidase
Number analyzed (Participants) | 1
kilograms
  Baseline | 2.5 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 5.8 (NA) — Standard deviation cannot be derived for a single participant.
  Week 24 | 7.8 (NA) — Standard deviation cannot be derived for a single participant.
  Week 36 | 9.2 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 9.9 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 | 10.8 (NA) — Standard deviation cannot be derived for a single participant.

25. Primary Outcome: Height of the Infant
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Laronidase
Number analyzed (Participants) | 1
centimeter
  Baseline | 50.0 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 64.0 (NA) — Standard deviation cannot be derived for a single participant.
  Week 24 | 66.5 (NA) — Standard deviation cannot be derived for a single participant.
  Week 36 | 72.0 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 76.5 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 | 78.0 (NA) — Standard deviation cannot be derived for a single participant.

26. Primary Outcome: Temperature of the Infant
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. Temperature was not measured at Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: Celcius
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Celcius
  Baseline: number analyzed (Participants) | 0
  Week 12: number analyzed (Participants) | 0
  Week 24 | 36.5 (NA) — Standard deviation cannot be derived for a single participant.
  Week 36 | 36.2 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 35.9 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 | 36.3 (NA) — Standard deviation cannot be derived for a single participant.

27. Primary Outcome: Head Circumference of the Infant
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Laronidase
Number analyzed (Participants) | 1
centimeter
  Baseline | 33 (NA) — Standard deviation cannot be derived for a single participant.
  Week 12 | 39 (NA) — Standard deviation cannot be derived for a single participant.
  Week 24 | 42 (NA) — Standard deviation cannot be derived for a single participant.
  Week 36 | 43.2 (NA) — Standard deviation cannot be derived for a single participant.
  Week 48 | 47 (NA) — Standard deviation cannot be derived for a single participant.
  Week 72 | 45 (NA) — Standard deviation cannot be derived for a single participant.

28. Primary Outcome: Number of Participants With Normal Overall Assessment Measured Using Denver II Developmental Screening Scores
Description: Infant development was assessed with the Denver II Developmental Screening Test. It consisted of 5 areas/subscore i.e., test behavior, personal-social, fine motor, language, and gross motor. The number of participants with normal overall assessment measured using Denver II Developmental Screening Scores have been reported by visit.
Time Frame: Week 12, Week 24, Week 36, Week 48, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants
  Week 12 | 1
  Week 24 | 1
  Week 36 | 1
  Week 48 | 1
  Week 72 | 1

29. Primary Outcome: Number of Infants With IgM and IgG Antibodies to Laronidase Present at Any Time Point
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase.
Measure: Count of Participants; unit: Participants
Arm/Group | Laronidase
Number analyzed (Participants) | 1
Participants
  IgG at Baseline | 1
  IgG at Week 12 | 0
  IgG at Week 24 | 0
  IgG at Week 36 | 0
  IgG at Week 72 | 0
  IgM at Baseline | 0
  IgM at Week 12 | 0
  IgM at Week 24 | 0
  IgM at Week 36 | 0
  IgM at Week 72 | 0

30. Primary Outcome: Time to Development of IgM and IgG Antibodies to Laronidase
Time Frame: up to Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. No IgM and IgG antibody was detected during the study, hence time is not-evaluable.
Arm/Group | Laronidase
Number analyzed (Participants) | 0

31. Primary Outcome: Amount of IgG and IgM Antibody Titers to Laronidase
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 72
Population: Infants who were breastfeed while the mothers were receiving laronidase. No IgG antibody was detected at Week 12, Week 24, Week 36, and Week 72. No IgM was detected at Baseline, Week 12, Week 24, Week 36, and Week 72.
Measure: Mean (Standard Deviation); unit: antibody titer
Arm/Group | Laronidase
Number analyzed (Participants) | 1
antibody titer
  IgG at Baseline | 6400 (NA) — Standard deviation cannot be derived for a single participant.
  IgG at Week 12: number analyzed (Participants) | 0
  IgG at Week 24: number analyzed (Participants) | 0
  IgG at Week 36: number analyzed (Participants) | 0
  IgG at Week 72: number analyzed (Participants) | 0
  IgM at Baseline: number analyzed (Participants) | 0
  IgM at Week 12: number analyzed (Participants) | 0
  IgM at Week 24: number analyzed (Participants) | 0
  IgM at Week 36: number analyzed (Participants) | 0
  IgM at Week 72: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 18 months for mother and 72 weeks for the infant.
Groups:
- Mothers Treated With Laronidase: Mothers treated with laronidase who intended to breastfeed their infants while receiving laronidase.
- Infants Who Were Breastfeed: Infants who were breastfeed while the mothers were receiving laronidase.
Arm/Group | Mothers Treated With Laronidase | Infants Who Were Breastfeed
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mothers Treated With Laronidase (N=1) | Infants Who Were Breastfeed (N=1)
Tachycardia (Cardiac disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Perinatal depression (Psychiatric disorders) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was conducted to fulfill a post marketing commitment (PMC). Upon acknowledgement of closure of PMC by FDA, the study was terminated by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-01-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT00418821/Prot_SAP_000.pdf